CLINICAL TRIAL: NCT03023930
Title: Opioid Use Disorder in the Emergency Department: Clinical Trials Network-0069
Brief Title: Opioid Use Disorder in the Emergency Department: CTN 0069
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1611018631; 5UG1DA015831-15 (NIH)
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Masking Description: Note: Care Providers and Research Associates are masked during Baseline Evaluation Period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evidenced-based Practice Dissemination (Experimental): Evaluating standard dissemination practice compared with implementation facilitation
  Interventions: Other: Standard Dissemination Practice; Other: Implementation Facilitation (IF)

INTERVENTIONS:
Other: Standard Dissemination Practice — Emergency department provider education using a grand rounds format. The content of the lecture will cover the scope of the opioid problem, ED specific facts related to the epidemic, potential models of intervention including the results of publications outlining the efficacy of ED-initiated BUP.
Other: Implementation Facilitation (IF) — IF involves a "formative evaluation" to identify the specific and dynamic needs of stakeholders and the context for implementation of evidence-based practices. This evaluation informs the initial tailoring and refinement of the IF, which includes a bundle of services tailored to meet site-specific needs, such as identifying and engaging local stakeholders, providing extensive ongoing education, tailoring program to the site and monitoring performance and offering feedback.

SUMMARY:
The purpose of this study is to evaluate the impact of (1) Implementation Facilitation (IF) on rates of provision of Emergency Department (ED)-initiated buprenorphine/naloxone (BUP) treatment with referral for ongoing medication-assisted treatment (MAT) and the (2) effectiveness of IF on patient engagement in formal addiction treatment at 30 days.

DETAILED DESCRIPTION:
The study was originally proposed to use a Hybrid Type 3 Effectiveness-Implementation framework and a modified stepped wedge design.

Original protocol registration language: The study will be conducted at four EDs with a high prevalence of patients with untreated opioid use disorder (OUD). The four sites will receive the same sequence of evaluations and interventions: the baseline evaluation period after the standard dissemination practice, the IF phase, and continuation of facilitation into the IF evaluation period. The timing of initiation of the study activities at each site will be randomly offset by ~ 3 month increments to accommodate logistical constraints of simultaneous implementation at all sites. The study populations will include (1) ED providers and staff involved in the treatment of patients with OUD; (2) Community opioid treatment provider and program staff involved in providing care for patients with OUD referred from the ED; and (3) ED patients with moderate to severe OUD.

Exploratory analyses have been added to assess the impact of COVID-19 and social distancing guidance on drug use and drug supply; access to medications for opioid use disorder; and COVID19 disease from the perspectives of patient participants and ED leadership.

Upon results entry, changes were made to reflect that the study design originally was described as a "modified step wedge" but ultimately was not designed or implemented as such, as there was no substantial overlap of the baseline evaluation and IF evaluation periods. Thus, the statistical plan was adjusted accordingly.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patients who are treated in the ED during study screening hours with Diagnostic and Statistical Manual (DSM)-5 criteria for moderate to severe OUD and provide an opioid positive urine sample will be eligible to participate.

Patient Exclusion Criteria:

* Patients who test positive for fentanyl only are not eligible due to lack of uniformly available rapid urine tests.
* Patients will be excluded if they have a medical or psychiatric condition requiring hospitalization at the index ED visit, are acutely suicidal or severely cognitively impaired precluding informed consent, present from an extended care facility, require continued prescription opioids for a pain condition, are a prisoner or in police custody at time of index ED visit, are currently (past 30 days) enrolled in formal addiction treatment including by court order, are unable to provide 2 contact numbers, are unwilling to follow study procedures, have been previously enrolled in the current study or do not speak English.

ED and Community Participants Inclusion Criteria:

* ED and community providers and administrators (i.e. physicians, residents, fellows, nursing, nurse practitioners, physician assistants, pharmacists, social workers, counselors, administrative directors, office-based physicians and opioid treatment program representatives) as well as ED patients with OUD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1731 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2022-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail D'Onofrio, MD, MS, Principal Investigator — Department of Emergency Medicine, Yale School of Medicine; David A Fiellin, MD, Principal Investigator — Department of Internal Medicine, Yale School of Medicine
Locations (5):
- United States (5):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Mount Sinai Hospital, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] D'Onofrio G, O'Connor PG, Pantalon MV, Chawarski MC, Busch SH, Owens PH, Bernstein SL, Fiellin DA. Emergency department-initiated buprenorphine/naloxone treatment for opioid dependence: a randomized clinical trial. JAMA. 2015 Apr 28;313(16):1636-44. doi: 10.1001/jama.2015.3474. PMID 25919527
- [Background] Coupet E Jr, D'Onofrio G, Chawarski M, Edelman EJ, O'Connor PG, Owens P, Martel S, Fiellin DA, Cowan E, Richardson L, Huntley K, Whiteside LK, Lyons MS, Rothman RE, Pantalon M, Hawk K. Emergency department patients with untreated opioid use disorder: A comparison of those seeking versus not seeking referral to substance use treatment. Drug Alcohol Depend. 2021 Feb 1;219:108428. doi: 10.1016/j.drugalcdep.2020.108428. Epub 2020 Nov 26. PMID 33307301
- [Background] Chawarski MC, Hawk K, Edelman EJ, O'Connor P, Owens P, Martel S, Coupet E Jr, Whiteside L, Tsui JI, Rothman R, Cowan E, Richardson L, Lyons MS, Fiellin DA, D'Onofrio G. Use of Amphetamine-Type Stimulants Among Emergency Department Patients With Untreated Opioid Use Disorder. Ann Emerg Med. 2020 Dec;76(6):782-787. doi: 10.1016/j.annemergmed.2020.06.046. Epub 2020 Aug 8. PMID 32782084
- [Background] Hawk KF, D'Onofrio G, Chawarski MC, O'Connor PG, Cowan E, Lyons MS, Richardson L, Rothman RE, Whiteside LK, Owens PH, Martel SH, Coupet E Jr, Pantalon M, Curry L, Fiellin DA, Edelman EJ. Barriers and Facilitators to Clinician Readiness to Provide Emergency Department-Initiated Buprenorphine. JAMA Netw Open. 2020 May 1;3(5):e204561. doi: 10.1001/jamanetworkopen.2020.4561. PMID 32391893
- [Background] D'Onofrio G, Edelman EJ, Hawk KF, Pantalon MV, Chawarski MC, Owens PH, Martel SH, VanVeldhuisen P, Oden N, Murphy SM, Huntley K, O'Connor PG, Fiellin DA. Implementation facilitation to promote emergency department-initiated buprenorphine for opioid use disorder: protocol for a hybrid type III effectiveness-implementation study (Project ED HEALTH). Implement Sci. 2019 May 7;14(1):48. doi: 10.1186/s13012-019-0891-5. PMID 31064390
- [Derived] D'Onofrio G, Edelman EJ, Hawk KF, Chawarski MC, Pantalon MV, Owens PH, Martel SH, Rothman R, Saheed M, Schwartz RP, Cowan E, Richardson L, Salsitz E, Lyons MS, Freiermuth C, Wilder C, Whiteside L, Tsui JI, Klein JW, Coupet E, O'Connor PG, Matthews AG, Murphy SM, Huntley K, Fiellin DA. Implementation Facilitation to Promote Emergency Department-Initiated Buprenorphine for Opioid Use Disorder. JAMA Netw Open. 2023 Apr 3;6(4):e235439. doi: 10.1001/jamanetworkopen.2023.5439. PMID 37017967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27,748 patients were screened during the baseline evaluation period and 394 were enrolled and analyzed. During the IF evaluation period, 26,456 were screened and 362 enrolled and analyzed. The study was originally conceived as a "modified step wedge" but not designed or implemented as such, as there was no substantial overlap of the baseline evaluation and IF evaluation periods. A total of 975 unique providers were assessed across the study periods via survey.
Groups:
- Baseline Evaluation Period Cohort; IF Evaluation Period: Evaluating standard dissemination practice compared with implementation facilitation
  Standard Dissemination Practice: Emergency department provider education using a grand rounds format. The content of the lecture will cover the scope of the opioid problem, ED specific facts related to the epidemic, potential models of intervention including the results of publications outlining the efficacy of ED-initiated BUP.
  Implementation Facilitation (IF): IF involves a "formative evaluation" to identify the specific and dynamic needs of stakeholders and the context for implementation of evidence-based practices. This evaluation informs the initial tailoring and refinement of the IF, which includes a bundle of services tailored to meet site-specific needs, such as identifying and engaging local stakeholders, providing extensive ongoing education, tailoring program to the site and monitoring performance and offering feedback.
- Providers - Baseline Period: Unique total number of providers added during Baseline Period
- Providers - 6 Month Period: Unique total number of providers added at 6 Month Period
- Providers - 12 Month Period: Unique total number of providers added at the 12 Month Period
Period: Overall Study
Arm/Group | Baseline Evaluation Period Cohort | IF Evaluation Period | Providers - Baseline Period | Providers - 6 Month Period | Providers - 12 Month Period
Started | 394 | 362 | 706 | 92 | 177
Completed | 394 | 362 | 706 | 92 | 177
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected for providers.
Groups:
- IF Evaluation Period Cohort: Evaluating standard dissemination practice compared with implementation facilitation
  Standard Dissemination Practice: Emergency department provider education using a grand rounds format. The content of the lecture will cover the scope of the opioid problem, ED specific facts related to the epidemic, potential models of intervention including the results of publications outlining the efficacy of ED-initiated BUP.
  Implementation Facilitation (IF): IF involves a "formative evaluation" to identify the specific and dynamic needs of stakeholders and the context for implementation of evidence-based practices. This evaluation informs the initial tailoring and refinement of the IF, which includes a bundle of services tailored to meet site-specific needs, such as identifying and engaging local stakeholders, providing extensive ongoing education, tailoring program to the site and monitoring performance and offering feedback.
- Total: Total of all reporting groups
Arm/Group | Baseline Evaluation Period Cohort | IF Evaluation Period Cohort | Total
Number analyzed (Participants) | 394 | 362 | 756
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (11.7) | 39.7 (11.7) | 39.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 95 | 216
  Male | 273 | 267 | 540
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 39 | 88
  Not Hispanic or Latino | 345 | 323 | 668
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 15 | 27
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 110 | 113 | 223
  White | 206 | 188 | 394
  More than one race | 14 | 16 | 30
  Unknown or Not Reported | 47 | 24 | 71
Region of Enrollment [Number; unit: participants]
  United States | 394 | 362 | 756
Education [Count of Participants; unit: Participants]
  Less than high school diploma | 140 | 126 | 266
  High school graduate or equivalent (GED) | 130 | 146 | 276
  Some college, no degree | 74 | 62 | 136
  ≥ College degree | 50 | 28 | 78
Employment [Count of Participants; unit: Participants]
  Working | 63 | 66 | 129
  Unemployed | 228 | 192 | 420
  Disabled permanently or temporarily | 80 | 62 | 142
Unstable Housing [Count of Participants; unit: Participants] — Spent at least one night in the past 12 months in any of the following places.
  Participants
    Shelter for homeless persons | 102 | 108 | 210
    On the street/public place not intended for sleeping | 191 | 192 | 383
    Doubled up in someone else's house apartment | 190 | 135 | 325
Currently living in any of the following places [Count of Participants; unit: Participants]
  Shelter for homeless persons | 41 | 41 | 82
  On the street or public place not intended for sleeping | 94 | 98 | 192
  Welfare hotel or SRO | 3 | 6 | 9
  Emergency, temporary, transitional or halfway house | 4 | 9 | 13
Health insurance [Count of Participants; unit: Participants]
  Private/commercial | 45 | 24 | 69
  Medicare | 31 | 37 | 68
  Medicaid | 287 | 254 | 541
  Unknown | 50 | 66 | 116
Primary Medical Provider [Count of Participants; unit: Participants] — Population: 393 out of 394 reported for Baseline Evaluation Period and 361 out of 362 reported for IF Evaluation Period
  Participants
    number analyzed (Participants) | 393 | 361 | 754
    Private physician office | 57 | 59 | 116
    Clinic | 116 | 96 | 212
    Emergency Department or none | 217 | 204 | 421
    Not reported | 3 | 2 | 5
Number of Positive UDS results by substance [Count of Participants; unit: Participants]
  Benzodiazepines | 101 | 126 | 227
  Amphetamine | 114 | 102 | 216
  Marijuana | 153 | 128 | 281
  Methamphetamine | 146 | 141 | 287
  Opiates (300 ng) | 328 | 283 | 611
  Cocaine | 177 | 165 | 342
  Ecstasy | 21 | 26 | 47
  Oxycodone | 159 | 139 | 298
  Methadone | 43 | 56 | 99
  Barbiturates | 7 | 1 | 8
  Buprenorphine | 144 | 169 | 313
  Fentanyl | 200 | 216 | 416
Overdose History [Count of Participants; unit: Participants]
  Overdosed at least once in the past 30 days | 108 | 106 | 214
  Report a medical intervention overdose | 84 | 79 | 163
  Injection drug use past month | 232 | 185 | 417
Mental Health History [Count of Participants; unit: Participants]
  Psych eval during the ED visit? | 11 | 15 | 26
  Lifetime psychiatric treatment: Inpatient | 161 | 116 | 277
  Lifetime psychiatric treatment: Outpatient | 185 | 150 | 335
  Any psychiatric treatment, past 30 day | 60 | 42 | 102

OUTCOME MEASURES:

1. Primary Outcome: Implementation (Considered the Primary Outcome)
Description: The primary implementation outcome will be evaluated assessing the rate of ED-initiated BUP therapy with referral for ongoing MAT
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Evaluation Period Cohort | IF Evaluation Period Cohort
Number analyzed (Participants) | 394 | 362
Participants | 2 | 53
Statistical Analysis 1: Comparison: Baseline Evaluation Period Cohort vs IF Evaluation Period Cohort; Test type: Superiority; p < 0.001, Regression, Logistic; proc logistic

2. Primary Outcome: Effectiveness
Description: The primary effectiveness outcome is defined as the rates of patient engagement in formal addiction treatment on the 30th day post enrollment.
Time Frame: 30 Days Post Enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Evaluation Period Cohort | IF Evaluation Period Cohort
Number analyzed (Participants) | 394 | 362
Participants | 40 | 59
Statistical Analysis 1: Comparison: Baseline Evaluation Period Cohort vs IF Evaluation Period Cohort; Test type: Superiority; p = 0.011, Regression, Logistic; proc logistic

3. Secondary Outcome: Implementation: ED Organizational Readiness to Change Assessment (ORCA) Score
Description: ED ORCA score relating to ED-initiated BUP with referral for ongoing MAT. Scores are dichotomized as less ready (scores 0-6) or most ready (scores 7-10).
Time Frame: Pre IF (Baseline)
Population: Clinicians assessed at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Evaluation Period Cohort
Number analyzed (Participants) | 268
Participants
  Most Ready | 56
  Less Ready | 212

4. Other Pre Specified Outcome: Implementation: ED Provider Readiness and Preparedness Ruler Score
Description: ED provider readiness and preparedness ruler score to initiate BUP and provide referral for ongoing MAT.
Time Frame: Pre IF (Baseline)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Implementation: ED Provider Readiness and Preparedness Ruler Score
Description: ED provider readiness and preparedness ruler score to initiate BUP and provide referral for ongoing MAT
Time Frame: post IF Evaluation Period (12 months)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Implementation: ED Provider Readiness and Preparedness Ruler Score
Description: ED provider readiness and preparedness ruler score to initiate BUP and provide referral for ongoing MAT
Time Frame: Post IF (6 months)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Effectiveness: Illicit Opioid Urine Toxicology
Description: Rates of illicit opioid negative urines
Time Frame: 30 days post enrollment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Effectiveness: Healthcare Service Utilization
Description: All Healthcare Service Utilization Inpatient and Outpatient
Time Frame: 30 days post enrollment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Effectiveness: Overdose Event
Description: Overdose event (past 30 days) captured by participant self-report, state medical examiner records, National Death Index and review of medical records
Time Frame: 30 days post enrollment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Effectiveness: Opioid Use
Description: Self-reported days of illicit opioid use (past 7 days) as measured by Time-Line Follow-Back methods at 30 days
Time Frame: 30 days post enrollment
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Effectiveness: HIV Risk
Description: HIV risk taking behaviors (past 30 days) as measured by HIV Risk Taking Behavior Scale
Time Frame: 30 days post enrollment
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Implementation: Community ORCA Score
Description: Community opioid treatment provider/program ORCA score relating to receiving patients with OUD who have received ED-initiated BUP
Time Frame: Pre IF (Baseline)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Implementation: Community ORCA Score
Description: as for outcome 12
Time Frame: Post IF (6 months)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Implementation: Community ORCA Score
Description: as for outcome 12
Time Frame: post IF Evaluation Period (12 months)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Implementation: Community Readiness and Preparedness Ruler Score
Description: Community opioid treatment provider/program readiness and preparedness ruler score to continue MAT for patients with OUD who have received ED-initiated BUP
Time Frame: Pre IF (Baseline)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Implementation: Community Readiness and Preparedness Ruler Score
Description: as for outcome 15
Time Frame: Post IF (6 months)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Implementation: Community Readiness and Preparedness Ruler Score
Description: as for outcome 15
Time Frame: post IF Evaluation Period (12 months)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Implementation: ED Organizational Readiness to Change Assessment (ORCA) Score
Description: ED ORCA score relating to ED-initiated BUP with referral for ongoing MAT
Time Frame: Post IF (6 months)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Implementation: ED Organizational Readiness to Change Assessment (ORCA) Score
Description: ED ORCA score relating to ED-initiated BUP with referral for ongoing MAT
Time Frame: Post IF Evaluation Period (12 months)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Implementation: Fidelity
Description: Fidelity will be measured using a critical action checklist relating to the provision of ED-initiated BUP with referral for ongoing MAT in eligible patients.
Time Frame: Baseline Period (Baseline)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Implementation: Fidelity
Description: as for outcome 20
Time Frame: IF Evaluation Period (18 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data was collected over 12 months.
Description: There was no adverse event monitoring for providers taking part in the study.
Arm/Group | Baseline Evaluation Period Cohort | IF Evaluation Period
All-Cause Mortality (participants affected / at risk) | 1/394 | 2/362
Serious Adverse Events (participants affected / at risk) | 0/394 | 0/362
Other Adverse Events (participants affected / at risk) | 0/394 | 0/362

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT03023930/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT03023930/SAP_001.pdf
  • Informed Consent Form (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03023930/ICF_002.pdf